CLINICAL TRIAL: NCT02572310
Title: A Prospective Radiostereometric Analysis (RSA) Study of Implant Stability and Clinical Evaluation of Simplex High Viscosity Bone Cement in Primary Total Knee Arthroplasty
Brief Title: Simplex High Viscosity Bone Cement in Primary Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael Dunbar (Other)
Responsible Party: Sponsor-Investigator, Michael Dunbar, Principal Investigator, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STR HVC
Record Dates: First submitted 2015-08-19; First posted 2015-10-08 (Estimated); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Osteoarthritis
Keywords: total knee arthroplasty
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HV Cement (Experimental): Simplex High Viscosity Bone Cement
  Interventions: Device: Simplex High Viscosity Bone Cement

INTERVENTIONS:
Device: Simplex High Viscosity Bone Cement — high viscosity bone cement for total knee replacement
  Other Names: HV Bone Cement

SUMMARY:
In this study the investigators propose to monitor subjects who have received Triathlon total knee components inserted with HV cement. The primary outcome will be fixation of the tibial implant component as assessed with RSA and to determine the functionality of patients after surgery using self-reported questionnaires. This is a historical control study, comparing the study cohort to a previous group with Triathlon implants and the long-standing Simplex T cement. The secondary outcomes are inducible displacements of the implants as well as a qualitative evaluation of the cement handling characteristics performed by the operating room staff.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic arthritis of the knee indicating primary total knee arthroplasty
* Between the ages of 21 and 80 inclusive
* Patients willing and able to comply with follow-up requirements and self-evaluations
* Ability to give informed consent

Exclusion Criteria:

* Active or prior infection
* Medical condition precluding major surgery
* Severe osteoporosis or osteopenia
* Neuromuscular impairment
* Significant co-morbidity affecting ability to ambulate

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-03; Primary Completion 2020-03 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Implant Migration measured with Radiostereometric Analysis (RSA) | 2 years
  Total implant migration will be measured in mm using RSA

SECONDARY OUTCOMES:
Qualitative handling characteristics captured through semi-structured interviews | intra-operative
  A qualitative methodology will be used to perform content analysis of the audio from the interviews stored in computer-assisted qualitative data analysis software. The content analysis will involve the use of a deductive approach to the interviews. The coding strategies will derived from a predetermined list of important qualities of bone cement and common themes will be identified as important for the usability of the new cement.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dunbar, PhD, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Nova Scotia Health Authority, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No
Local ethics approval does not permit sharing of individual participant data